CLINICAL TRIAL: NCT00292227
Title: Double-blind, Randomized, Placebo- and Positive-controlled, Parallel-group Trial to Assess the Potential Electrocardiographic Effects of Rotigotine Transdermal System up to 120 cm2/54.0 mg/Day in Subjects With Advanced-stage Idiopathic Parkinson's Disease: A Thorough QT/QTc Trial.
Brief Title: Cardiac Effects of Rotigotine Transdermal System in Subjects With Advanced-stage Idiopathic Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0864
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: advanced-stage idiopathic Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine Patch
  Interventions: Drug: Rotigotine; Other: Placebo infusion
- Placebo (Placebo Comparator): Placebo patch
  Interventions: Other: Placebo; Drug: Moxifloxacin infusion; Other: Placebo infusion

INTERVENTIONS:
Drug: Rotigotine — Rotigotine patch applied once daily for a 24-hour period.
  Rotigotine dose schedule (patch application days):
  Day 1 through Day 7: 9.0 mg/day; Day 8 through Day 14: 18.0 mg/day; Day 15 through Day 21: 27.0 mg/day; Day 22 through Day 28: 36.0 mg/day; Day 29 through Day 35: 45.0 mg/day; Day 36 through Day 42: 54.0 mg/day; Day 43 through Day 44: 45.0 mg/day; Day 45 through Day 46: 36.0 mg/day; Day 47 through Day 48: 27.0 mg/day; Day 49 through Day 50: 18.0 mg/day; Day 51 through Day 52: 9.0 mg/day;
  Other Names: Neupro
  Arms: Rotigotine
Other: Placebo — Placebo patch applied once daily for a 24-hour period. Size and number of patches matching to rotigotine dose schedule (patch application days):
  Day 1 through Day 7: 9.0 mg/day; Day 8 through Day 14: 18.0 mg/day; Day 15 through Day 21: 27.0 mg/day; Day 22 through Day 28: 36.0 mg/day; Day 29 through Day 35: 45.0 mg/day; Day 36 through Day 42: 54.0 mg/day; Day 43 through Day 44: 45.0 mg/day; Day 45 through Day 46: 36.0 mg/day; Day 47 through Day 48: 27.0 mg/day; Day 49 through Day 50: 18.0 mg/day; Day 51 through Day 52: 9.0 mg/day;
  Arms: Placebo
Drug: Moxifloxacin infusion — Moxifloxacin 400 mg/250 mL iv solution infused over 1h once either on Day 32 or on Day 39
  Arms: Placebo
Other: Placebo infusion — Placebo saline solution 250 mL infused over 1h once either on Day 32 or on Day 39
  Arms: Placebo
Other: Placebo infusion — Placebo saline solution 250 mL infused over 1h once on both Day 32 and on Day 39
  Arms: Rotigotine

SUMMARY:
The purpose of this trial is to assess whether rotigotine has an effect on the electrical activity of the heart. Moxifloxacin infusion is used as positive control to assess assay sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Advanced-stage idiopathic Parkinson's disease requiring treatment with levodopa.
* Nonchildbearing potential

Exclusion Criteria:

* Atypical Parkinson's syndrome(s).
* History of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant.
* Significant tremor or dyskinesias.
* Severe dysfunction of the autonomic nervous system.
* History of transient ischemic attack or stroke within the last 12 months.
* Conduction abnormality or relevant cardiac dysfunction and/or myocardial infarction within last 12 months.
* History or current condition of additional risk factors for Torsade de Pointes (eg, heart failure, hypokalemia), or a family history of long QT syndrome and/or of Torsade de Pointes.
* No stable sinus rhythm: more than 20 ectopics/h.
* Any other clinically relevant ECG abnormality.
* History or current condition of epilepsy and/or seizures.
* History or current condition of atopic or eczematous dermatitis, psoriasis, or another active skin disease.
* History or current condition of symptomatic orthostatic hypotension.
* History or current condition of significant skin hypersensitivity to adhesives or other transdermal products or recent unresolved contact dermatitis.
* History of glucose 6-phosphate dehydrogenase deficiency.
* History of tendonitis or tendon rupture with quinolone antibiotics.
* Renal or hepatic dysfunction.
* Treatment with dopamine agonists, MAO A inhibitors, reserpine, or alpha-methyldopa
* Therapy known to produce a nontrivial prolongation of the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (2):
- South Africa (2):
  - Farmovs-Parexel (Pty) Ltd, Bloemfontein
  - Qdot, a division of Parexel International DA (Pty) Ltd., George

REFERENCES:
- [Result] Malik M, Andreas JO, Hnatkova K, Hoeckendorff J, Cawello W, Middle M, Horstmann R, Braun M. Thorough QT/QTc study in patients with advanced Parkinson's disease: cardiac safety of rotigotine. Clin Pharmacol Ther. 2008 Nov;84(5):595-603. doi: 10.1038/clpt.2008.143. Epub 2008 Jul 23. PMID 18650802
- [Result] Elshoff JP, Braun M, Andreas JO, Middle M, Cawello W. Steady-state plasma concentration profile of transdermal rotigotine: an integrated analysis of three, open-label, randomized, phase I multiple dose studies. Clin Ther. 2012 Apr;34(4):966-78. doi: 10.1016/j.clinthera.2012.02.008. Epub 2012 Mar 7. PMID 22401642
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Within the placebo patch group, subjects were randomized to the sequence of receiving either placebo saline iv solution or moxifloxacin iv solution on Days 32 and 39 in a cross-over design. This treatment was in addition to treatment with the placebo patch. Subjects in the rotigotine patch group received placebo iv solution on Day 32 and Day 39.
Groups:
- Rotigotine Patch (Infusion: Placebo-Placebo): Rotigotine Patch applied once daily for a 24 hour period over a total period of 52 days following the prespecified dosing schedule. Placebo saline solution 250 mL infused over 1 hour on Day 32 and on Day 39.
- Placebo Patch (Infusion: Moxifloxacin-Placebo): Placebo Patch applied once daily for a 24 hour period over a total period of 52 days following the prespecified dosing schedule. Moxifloxacin 400 mg/250 mL iv solution infused over 1 hour on Day 32. Placebo saline solution 250 mL infused over 1 hour on Day 39.
- Placebo Patch (Infusion: Placebo-Moxifloxacin): Placebo Patch applied once daily for a 24 hour period over a total period of 52 days following the prespecified dosing schedule. Placebo saline solution 250 mL infused over 1 hour on Day 32. Moxifloxacin 400 mg/250 mL iv solution infused over 1 hour on Day 39.
Period: Patch Period
Arm/Group | Rotigotine Patch (Infusion: Placebo-Placebo) | Placebo Patch (Infusion: Moxifloxacin-Placebo) | Placebo Patch (Infusion: Placebo-Moxifloxacin)
Started | 66 | 31 | 33
Completed | 65 | 31 | 30
Not Completed | 1 | 0 | 3
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Cross-over Period 1 (Day 32)
Arm/Group | Rotigotine Patch (Infusion: Placebo-Placebo) | Placebo Patch (Infusion: Moxifloxacin-Placebo) | Placebo Patch (Infusion: Placebo-Moxifloxacin)
Started | 65 | 31 | 30
Completed | 65 | 31 | 30
Not Completed | 0 | 0 | 0
Period: Cross-over Period 2 (Day 39)
Arm/Group | Rotigotine Patch (Infusion: Placebo-Placebo) | Placebo Patch (Infusion: Moxifloxacin-Placebo) | Placebo Patch (Infusion: Placebo-Moxifloxacin)
Started | 65 | 31 | 30
Completed | 65 | 31 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rotigotine Patch: Rotigotine Patch applied once daily for a 24 hour period over a total period of 52 days following the prespecified dosing schedule.
- Placebo Patch: Placebo patch applied once daily for a 24 hour period over a total period of 52 days following the prespecified dosing schedule.
- Total: Total of all reporting groups
Arm/Group | Rotigotine Patch | Placebo Patch | Total
Number analyzed (Participants) | 66 | 64 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 36 | 29 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.4) | 63.1 (9.8) | 63.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 45 | 44 | 89
Region of Enrollment [Number; unit: participants]
  South Africa | 66 | 64 | 130

OUTCOME MEASURES:

1. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI at Time of Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 20:00h.
Time Frame: Baseline (Day -2/ Day -1) 20:00h, Day 42 20:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 0.46 (5.96) | 1.13 (6.86)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; The analysis was based on a non-inferiority comparison of rotigotine vs placebo using a 1-sided 95% confidence interval (or, equivalently, the upper limit of 2-sided 90% confidence interval) for the time-matched changes from Baseline in QTcI; Test type: Non-Inferiority or Equivalence — A standard deviation of 12ms was assumed for sample size calculation. Sample size was calculated to have 90% power to show the non-inferiority of rotigotine against placebo with respect to the non-inferiority margin of 10ms (α=0.05, 1-sided); ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.75, 90% CI [-2.63 to 1.12] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

2. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 1 Hour After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 21:00h.
Time Frame: Baseline (Day -2/ Day -1) 21:00h, Day 42 21:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.82 (8.32) | 1.67 (7.25)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.01, 90% CI [-2.21 to 2.19] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

3. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 2 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 22:00h.
Time Frame: Baseline (Day -2/ Day -1) 22:00h, Day 42 22:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 64 | 61
milliseconds [ms] | 2.55 (6.96) | 1.78 (6.76)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.84, 90% CI [-1.12 to 2.80] — The direction of the estimate is Rotigotine - Placebo Mean difference was estimated from the ANCOVA model

4. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 3 Hours After Patch Application on Day 42(Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 23:00h.
Time Frame: Baseline (Day -2/ Day -1) 23:00h, Day 42 23:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.02 (7.98) | 0.89 (6.52)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.26, 90% CI [-1.80 to 2.32] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

5. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 4 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 00:00h.
Time Frame: Baseline (Day -2/ Day -1) 00:00h, Day 43 00:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 0.54 (8.09) | 0.83 (7.29)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.11, 90% CI [-2.25 to 2.02] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

6. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 5 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 1:00h.
Time Frame: Baseline (Day -2/ Day -1) 1:00h, Day 43 1:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.17 (7.97) | 0.03 (8.11)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.07, 90% CI [-2.14 to 2.28] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

7. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 6 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 2:00h.
Time Frame: Baseline (Day -2/ Day -1) 2:00h, Day 43 2:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 64 | 61
milliseconds [ms] | -0.62 (8.57) | 0.05 (7.39)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.56, 90% CI [-2.84 to 1.72] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

8. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 7 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 3:00h.
Time Frame: Baseline (Day -2/ Day -1) 3:00h, Day 43 3:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.63 (7.84) | -0.26 (6.44)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.26, 90% CI [-2.29 to 1.78] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

9. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 8 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 4:00h.
Time Frame: Baseline (Day -2/ Day -1) 4:00h, Day 43 4:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.31 (8.41) | 0.95 (5.75)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -1.17, 90% CI [-3.25 to 0.91] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

10. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 9 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 5:00h.
Time Frame: Baseline (Day -2/ Day -1) 5:00h, Day 43 5:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.39 (7.10) | -1.97 (7.12)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 1.69, 90% CI [-0.34 to 3.73] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

11. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 10 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 6:00h.
Time Frame: Baseline (Day -2/ Day -1) 6:00h, Day 43 6:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 63 | 61
milliseconds [ms] | 0.92 (7.70) | 0.58 (6.52)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.31, 90% CI [-1.70 to 2.32] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

12. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 11 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 7:00h.
Time Frame: Baseline (Day -2/ Day -1) 7:00h, Day 43 7:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 62 | 60
milliseconds [ms] | 1.94 (9.64) | 0.30 (5.90)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 1.65, 90% CI [-0.65 to 3.96] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

13. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 12 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 8:00h.
Time Frame: Baseline (Day -2/ Day -1) 8:00h, Day 43 8:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.16 (5.65) | 1.31 (5.26)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.21, 90% CI [-1.78 to 1.36] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

14. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 13 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 9:00h.
Time Frame: Baseline (Day -2/ Day -1) 9:00h, Day 43 9:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 0.83 (6.70) | 1.40 (5.78)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.53, 90% CI [-2.37 to 1.30] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

15. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 14 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 10:00h.
Time Frame: Baseline (Day -2/ Day -1) 10:00h, Day 43 10:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 64 | 61
milliseconds [ms] | 1.83 (6.96) | 2.12 (6.01)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.41, 90% CI [-2.30 to 1.49] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

16. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 15 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 11:00h.
Time Frame: Baseline (Day -2/ Day -1) 11:00h, Day 43 11:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.15 (6.42) | 1.60 (6.21)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.50, 90% CI [-2.34 to 1.35] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

17. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 16 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 12:00h.
Time Frame: Baseline (Day -2/ Day -1) 12:00h, Day 43 12:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 2.21 (6.96) | 1.99 (6.46)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.21, 90% CI [-1.76 to 2.17] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

18. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 17 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 13:00h.
Time Frame: Baseline (Day -2/ Day -1) 13:00h, Day 43 13:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.35 (6.10) | 2.59 (5.82)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -1.23, 90% CI [-2.99 to 0.53] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

19. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 18 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 14:00h.
Time Frame: Baseline (Day -2/ Day -1) 14:00h, Day 43 14:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 63 | 60
milliseconds [ms] | -0.31 (8.48) | 1.29 (6.43)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -1.62, 90% CI [-3.87 to 0.63] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

20. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 19 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 15:00h.
Time Frame: Baseline (Day -2/ Day -1) 15:00h, Day 43 15:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 64 | 61
milliseconds [ms] | 0.71 (6.01) | 1.51 (5.65)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.81, 90% CI [-2.55 to 0.93] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

21. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 20 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 16:00h.
Time Frame: Baseline (Day -2/ Day -1) 16:00h, Day 43 16:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.58 (6.07) | 1.90 (5.95)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.37, 90% CI [-2.13 to 1.39] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

22. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 21 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 17:00h.
Time Frame: Baseline (Day -2/ Day -1) 17:00h, Day 43 17:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.13 (6.92) | 0.57 (6.06)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.68, 90% CI [-2.60 to 1.25] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

23. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 22 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 18:00h.
Time Frame: Baseline (Day -2/ Day -1) 18:00h, Day 43 18:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.45 (6.60) | 0.27 (6.08)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 1.17, 90% CI [-0.69 to 3.03] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

24. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 23 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: Change in QTcI was analyzed by a parallel-group comparison between rotigotine patch and placebo patch. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). The baseline QTcI value was obtained from the average of the ECG assessment on Day -2 and Day -1. Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 19:00h.
Time Frame: Baseline (Day -2/ Day -1) 19:00h, Day 43 19:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | 1.50 (6.70) | 0.64 (6.43)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = 0.80, 90% CI [-1.14 to 2.73] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

25. Primary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTc Based on the QTcI 24 Hours After Patch Application on Day 42 (Rotigotine Dose of 54 mg/Day) (Parallel-group Comparison)
Description: as for outcome 1
Time Frame: Baseline (Day -2/ Day -1) 20:00h, Day 43 20:00h
Population: Safety population; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Rotigotine Patch | Placebo Patch
Number analyzed (Participants) | 65 | 61
milliseconds [ms] | -0.96 (7.08) | -0.58 (5.79)
Statistical Analysis 1: Comparison: Rotigotine Patch vs Placebo Patch; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; The ANCOVA model included the factors site, treatment, gender, and time-matched baseline QTcI as covariate; Mean Difference (Net) = -0.42, 90% CI [-2.33 to 1.50] — The direction of the estimate is Rotigotine - Placebo. Mean difference was estimated from the ANCOVA model

26. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 2 Hours Before Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 8:00h.
Time Frame: Baseline (Day -2/ Day -1) 8:00h, Day 32/ Day 39 8:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Groups:
- Moxifloxacin Infusion: Moxifloxacin 400 mg/250 mL iv solution infused over 1 hour once either on Day 32 or on Day 39.
- Placebo Infusion: Placebo saline solution 250 mL infused over 1 hour once either on Day 32 or on Day 39.
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 60
milliseconds [ms] | 1.70 (5.76) | 1.29 (6.48)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; For the analysis of the assay sensitivity, an ANOVA with the factors treatment, period, sequence, and subject(sequence) for comparison of moxifloxacin vs placebo (cross-over comparison) was performed. The point estimates for the difference between placebo and positive control (moxifloxacin) and the respective 95% confidence intervals were calculated; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 0.34, 95% CI [-1.04 to 1.71] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

27. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 1 Hour Before Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 9:00h.
Time Frame: Baseline (Day -2/ Day -1) 9:00h, Day 32/ Day 39 9:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 1.84 (5.97) | 1.36 (6.03)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 0.48, 95% CI [-0.72 to 1.68] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

28. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI at Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 10:00h.
Time Frame: Baseline (Day -2/ Day -1) 10:00h, Day 32/ Day 39 10:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 60
milliseconds [ms] | 2.21 (6.19) | 0.82 (7.34)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 1.51, 95% CI [0.30 to 2.73] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

29. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 1 Hour After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 11:00h.
Time Frame: Baseline (Day -2/ Day -1) 11:00h, Day 32/ Day 39 11:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 17.19 (7.49) | 3.70 (5.72)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 13.50, 95% CI [11.78 to 15.22] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

30. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 2 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 12:00h.
Time Frame: Baseline (Day -2/ Day -1) 12:00h, Day 32/ Day 39 12:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 12.44 (7.94) | 1.42 (6.08)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 11.02, 95% CI [9.12 to 12.93] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

31. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 3 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 13:00h.
Time Frame: Baseline (Day -2/ Day -1) 13:00h, Day 32/ Day 39 13:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 60 | 61
milliseconds [ms] | 12.68 (7.35) | 1.44 (5.91)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 11.30, 95% CI [9.94 to 12.67] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

32. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 4 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 14:00h.
Time Frame: Baseline (Day -2/ Day -1) 14:00h, Day 32/ Day 39 14:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 60
milliseconds [ms] | 9.48 (6.95) | 1.28 (6.37)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 8.28, 95% CI [6.85 to 9.70] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

33. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 5 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 15:00h.
Time Frame: Baseline (Day -2/ Day -1) 15:00h, Day 32/ Day 39 15:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 60
milliseconds [ms] | 10.06 (6.53) | 0.08 (5.50)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 9.30, 95% CI [7.57 to 11.02] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

34. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 6 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 16:00h.
Time Frame: Baseline (Day -2/ Day -1) 16:00h, Day 32/ Day 39 16:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 9.98 (6.74) | 1.10 (4.93)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 8.87, 95% CI [7.47 to 10.28] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

35. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 7 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 17:00h.
Time Frame: Baseline (Day -2/ Day -1) 17:00h, Day 32/ Day 39 17:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 8.97 (6.47) | 0.37 (6.14)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 8.60, 95% CI [7.25 to 9.96] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

36. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 8 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 18:00h.
Time Frame: Baseline (Day -2/ Day -1) 18:00h, Day 32/ Day 39 18:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 7.74 (5.84) | 0.22 (5.14)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 7.52, 95% CI [6.31 to 8.72] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

37. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 9 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 19:00h.
Time Frame: Baseline (Day -2/ Day -1) 19:00h, Day 32/ Day 39 19:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 7.33 (6.26) | -0.25 (5.51)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 7.58, 95% CI [6.21 to 8.95] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

38. Secondary Outcome: Time-matched Change From Baseline (Average of Day -2 and Day -1) in QTcI 10 Hours After Start of Infusion on Day 32 or Day 39 (Positive Control) and Respective Day 39 or Day 32 (Corresponding Placebo) (Cross-over Comparison)
Description: Change in QTcI was analyzed by a cross-over comparison between moxifloxacin infusion and placebo infusion. The QT interval refers to the respective time interval in the Electrocardiogram (ECG). The QT interval was corrected for heart rate using an individualized heart rate correction formula including QT/RR curvature optimization (QTcI). Absolute values are presented as unadjusted Mean and Standard Deviation. Baseline and final measures were taken at 20:00h.
Time Frame: Baseline (Day -2/ Day -1) 20:00h, Day 32/ Day 39 20:00h
Population: Safety population within the placebo patch group; only non-missing values were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds [ms]
Arm/Group | Moxifloxacin Infusion | Placebo Infusion
Number analyzed (Participants) | 61 | 61
milliseconds [ms] | 6.34 (6.13) | 0.14 (4.98)
Statistical Analysis 1: Comparison: Moxifloxacin Infusion vs Placebo Infusion; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; ANOVA; The ANOVA model included the factors treatment, period, sequence, and subject(sequence); Mean Difference (Net) = 6.19, 95% CI [4.94 to 7.45] — The direction of the estimate is Moxifloxacin - Placebo. Mean difference was estimated from the ANOVA model

ADVERSE EVENTS:
Time Frame: Adverse events are reported for the whole study period including the adverse events that occured during moxifloxacin or placebo infusion on day 32 or day 39.
Arm/Group | Rotigotine Patch | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/64
Other Adverse Events (participants affected / at risk) | 63/66 | 54/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine Patch (N=66) | Placebo Patch (N=64)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine Patch (N=66) | Placebo Patch (N=64)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Meniere's Disease (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Visual Disturbance (Eye disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 28 (71) | 14 (16)
Vomiting (Gastrointestinal disorders) | 15 (26) | 3 (4)
Lip Dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application Site Irritation (General disorders) | 3 (3) | 1 (1)
Application Site Oedema (General disorders) | 1 (1) | 0 (0)
Application Site Pruritus (General disorders) | 6 (7) | 2 (2)
Application Site Reaction (General disorders) | 3 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 3 (5)
Infusion Related Reaction (General disorders) | 0 (0) | 1 (1)
Infusion Site Pruritus (General disorders) | 0 (0) | 1 (1)
Infusion Site Reaction (General disorders) | 0 (0) | 1 (1)
Injection Site Thrombosis (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (3)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Tinea Cruris (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Failure Of Implant (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical Device Site Reaction (Injury, poisoning and procedural complications) | 15 (17) | 14 (16)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail Avulsion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Potassium Increased (Investigations) | 2 (2) | 1 (1)
Serum Ferritin Decreased (Investigations) | 0 (0) | 1 (1)
Serum Ferritin Increased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Balance Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 3 (3) | 1 (1)
Syncope Vasovagal (Nervous system disorders) | 2 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 5 (7) | 2 (3)
Headache (Nervous system disorders) | 19 (30) | 16 (27)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 19 (29) | 6 (6)
Paraesthesia (Nervous system disorders) | 1 (1) | 2 (2)
Parkinson's Disease (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (3)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (3) | 1 (1)
Disorientation (Psychiatric disorders) | 2 (4) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bruxism (Psychiatric disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Varicose Vein (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic Hypotension (Vascular disorders) | 5 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.